CLINICAL TRIAL: NCT02754557
Title: Physiological Augmentation of Mindfulness Meditation
Acronym: PAMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Negar Fani, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00085711
Record Dates: First submitted 2016-04-06; First posted 2016-04-28 (Estimated); Results first posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-09

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Trauma; PTSD; Mindfulness; Meditation; Neuroimaging; MRI
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Breath-Focused Meditation (Experimental): Women with post traumatic stress disorder (PTSD) will receive breath-focused meditation.
  Interventions: Other: Breath-Focused Meditation
- Breath-Focused Meditation + Physiological Feedback (Experimental): Women with post traumatic stress disorder (PTSD) will receive breath-focused meditation and physiological feedback.
  Interventions: Other: Breath-Focused Meditation; Device: Physiological Feedback

INTERVENTIONS:
Other: Breath-Focused Meditation — Participants will attend two breath-focused meditation sessions per week for three weeks. During the breath focus task, participants are asked to alternatively focus their breathing (1.5 minutes of breathing and 15 seconds of rest). Participants will be asked to "attend to the changing patterns of physical sensations as the breath moves in and out of your body. Focus your awareness on any sensations you may experience (e.g., your abdominal wall rising). Follow the sensations as you breathe in and all the way through until your breath leaves your body".
Device: Physiological Feedback — Participants will receive breath feedback, via dynamic velocity estimates from a respiration belt, which allows an analog of breath to be felt as vibration on their wrist via a tactile transducer on a table. The transducer is tuned to produce low frequencies so there is more vibration and less of an audible component than a regular speaker would produce.
  Arms: Breath-Focused Meditation + Physiological Feedback

SUMMARY:
The purpose of the study is to compare the efficacy of a physiologically-augmented breath-focused mindfulness-based intervention to reduce symptoms of dissociation that are associated with psychological trauma, as well as symptoms of posttraumatic stress disorder (PTSD). The study will evaluate whether physiological augmentation produces a greater change in dissociative symptoms, meditative engagement and attentional control, compared to non-augmented mindfulness. The augmentation comprises physiological feedback in the form of a vibration on the wrist. Vibrations are delivered by a device that will be placed on a participant's arm; the device vibrates in proportion to the person's breath.

DETAILED DESCRIPTION:
Chronically traumatized people are at much higher risk for developing dissociative symptoms, which are notoriously difficult to treat, particularly in the context of other posttraumatic stress disorder symptoms. Dissociation is a phenomenon that involves feelings of separation from one's body and emotional state. Mindfulness practices, including breath-focused mindfulness meditation, are known to be useful for improving attention to one's physiological state, thus enhancing a feeling of "connection" with one's present experience. However, mindfulness-based practices are naturally a challenging task for highly dissociative people. The present project proposes the use of a novel device that uses physiological feedback to boost the effects of breath-focused mindfulness meditation in this population. This device is an element placed on the wrist that vibrates in accordance with one's breath. The method capitalizes on a "bottom-up" neurophysiological process. This study plans to recruit 80 highly dissociative traumatized African American women through an established and highly productive NIH-funded project. Participants will be randomly assigned to 6 sessions of either breath-focused mindfulness meditation or physiologically augmented breath-focused mindfulness meditation. Electroencephalography data will be collected during the intervention sessions, and functional magnetic resonance imaging data will be collected pre- and post-intervention. These methods will be used to assess whether the physiological augmentation is producing: increased coherence or "network-like" activity among brain regions involved with interoception (awareness of one's bodily state); selective attention to the breath (increased temporo-parietal EEG gamma) and meditative engagement (increased frontal EEG theta). Clinical and neuropsychological measures will be used to assess potential effects on dissociative and posttraumatic symptoms, as well as selective and sustained attention and mindfulness ability. A follow-up will be conducted 1 month post-treatment to examine sustained clinical and cognitive effects.

ELIGIBILITY:
Inclusion Criteria:

* Experience of at least one Criterion A trauma
* Presence of current symptoms of post traumatic stress disorder (PTSD) that are significantly interfering with functioning
* Multiscale Dissociation Inventory depersonalization score of 7
* Fulfill at least two of the Clinician Administered PTSD Subscale criteria of clinically significant re-experiencing, avoidance, alterations in mood and cognitions, hyperarousal
* Willingness to participate in the study

Exclusion Criteria:

* Actively psychotic
* Cognitively compromised
* Pregnancy
* Substance or Alcohol Dependence

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Negar Fani, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Health System, Atlanta, Georgia
  - Wesley Woods Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Powers A, Dixon HD, Guelfo A, Mekawi Y, Bradley B, Kaslow N, Fani N. The mediating role of emotion dysregulation in the association between trait mindfulness and PTSD symptoms among trauma-exposed adults. Mindfulness (N Y). 2021 Sep;12(9):2229-2240. doi: 10.1007/s12671-021-01684-8. Epub 2021 Jul 16. PMID 34603539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Grady Memorial Hospital and the Wesley Woods Center in Atlanta, Georgia, USA. Participant enrollment began in March 2016 and the one month follow-up assessments were completed by September 21, 2021.
Groups:
- Breath-Focused Meditation: Women with post traumatic stress disorder receiving breath-focused meditation
- Breath-Focused Meditation Plus Physiological Feedback: Women with post traumatic stress disorder receiving breath-focused meditation augmented with physiological feedback
Period: Overall Study
Arm/Group | Breath-Focused Meditation | Breath-Focused Meditation Plus Physiological Feedback
Started | 27 | 38
Completed Post-treatment Assessment at Week 4 | 27 | 38
Completed One-month Post-treatment Assessment at Week 8 | 19 | 32
Completed (Completed the primary aim of the study which was the post-treatment follow up assessment at Week 4.) | 27 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Breath-Focused Meditation | Breath-Focused Meditation Plus Physiological Feedback | Total
Number analyzed (Participants) | 27 | 38 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.48 (11.97) | 40.11 (12.22) | 42.38 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 38 | 65
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 27 | 36 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 23 | 30 | 53
  White | 3 | 4 | 7
  More than one race | 1 | 1 | 2
  Other | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 38 | 65

OUTCOME MEASURES:

1. Primary Outcome: Multiscale Dissociation Inventory (MDI) Score
Description: The MDI is a 30-item self-report test of dissociative symptomology and it measures six different types of dissociative response. The scales of the MDI are disengagement, depersonalization, derealization, emotional constriction/numbing, memory disturbance, identity dissociation, and total dissociation. Items are scored from 1 to 5 where 1 = never and 5 = very often. Total scores range from 30 to 150 where higher scores indicate greater symptoms of dissociation.
Time Frame: Baseline, Week 4 (post-treatment), Week 8 (one month post-treatment)
Population: This analysis includes participants who attended the indicated study visit. One participant in the Breath-Focused Meditation Plus Physiological Feedback group attended the one month post-treatment visit but did not complete the MDI.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breath-Focused Meditation | Breath-Focused Meditation Plus Physiological Feedback
Number analyzed (Participants) | 27 | 38
score on a scale
  Baseline | 53.19 (12.99) | 61.58 (20.00)
  Post-treatment (Week 4) | 47.15 (15.13) | 51.00 (15.53)
  One Month Post-Treatment (Week 8): number analyzed (Participants) | 19 | 31
  One Month Post-Treatment (Week 8) | 44.11 (14.44) | 47.94 (17.82)

2. Primary Outcome: Modified PTSD Symptom Scale (MPSS) Score
Description: The MPSS is an 18-item instrument assessing the presence and severity of PTSD symptoms related to specific traumatic events in individuals with a known trauma history. Respondents indicate how frequently they experience each item on a scale of 0 to 3 where 0 = not at all and 3 = almost always. PTSD symptomatology over the prior 2 weeks is assessed, yielding a continuous measure of PTSD symptom severity ranging from 0 to 54. A higher score indicates greater symptom severity.
Time Frame: Baseline, Week 4 (post-treatment), Week 8 (one month post-treatment)
Population: This analysis includes participants who attended the indicated study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breath-Focused Meditation | Breath-Focused Meditation Plus Physiological Feedback
Number analyzed (Participants) | 27 | 38
score on a scale
  Baseline | 27.33 (7.23) | 28.82 (8.37)
  Post-treatment (Week 4) | 19.63 (10.54) | 20.97 (12.27)
  One Month Post-treatment (Week 8): number analyzed (Participants) | 19 | 32
  One Month Post-treatment (Week 8) | 17.58 (10.52) | 19.44 (12.69)

3. Primary Outcome: Kentucky Mindfulness Scale Score
Description: The Kentucky Mindfulness Scale is a 39-item scale that assesses skills related to what one does while practicing mindfulness. Items are rated on a 5 point Likert scale ranging from 1 (never or very rarely true) to 5 (almost always or always true). Items reflect either direct descriptions of the mindfulness skills, or they describe the absence of that skill and are reverse scored. Total scores range from 39 to 195 and higher scores reflect more mindfulness.
Time Frame: Baseline, Week 4 (post-treatment), Week 8 (one month post-treatment)
Population: This analysis includes participants who attended the indicated study visit. One participant in the Breath-Focused Meditation Plus Physiological Feedback group attended the one month post-treatment visit but did not complete the Kentucky Mindfulness Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breath-Focused Meditation | Breath-Focused Meditation Plus Physiological Feedback
Number analyzed (Participants) | 27 | 38
score on a scale
  Baseline | 122.19 (17.68) | 117.55 (19.24)
  Post-treatment (Week 4) | 125.37 (20.25) | 125.79 (17.29)
  One Month Post-treatment (Week 8): number analyzed (Participants) | 19 | 31
  One Month Post-treatment (Week 8) | 124.58 (22.25) | 126.65 (16.78)

4. Primary Outcome: Multidimensional Assessment of Interoceptive Awareness Score
Description: This is a clinical measure that assesses various aspects of interoception, including ability to attend to body sensations, regulate distress by attending to body sensations, and experiencing body sensations as safe and trustworthy. The instrument includes 32 items and which are scored from 0 to 5, where 0 = never and 5 = always. Total scores range from 0 to 160 and higher scores indicate greater awareness of body sensations.
Time Frame: Baseline, Week 4 (post-treatment), Week 8 (one month post-treatment)
Population: This analysis includes participants who attended the indicated study visit. One participant in the Breath-Focused Meditation Plus Physiological Feedback group attended the one month post-treatment visit but did not complete the Multidimensional Assessment of Interoceptive Awareness assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breath-Focused Meditation | Breath-Focused Meditation Plus Physiological Feedback
Number analyzed (Participants) | 27 | 38
score on a scale
  Baseline | 98.22 (24.39) | 86.45 (25.03)
  Post-treatment (Week 4) | 107.37 (31.46) | 106.92 (24.94)
  One Month Post-treatment (Week 8): number analyzed (Participants) | 19 | 31
  One Month Post-treatment (Week 8) | 110.63 (28.29) | 105.29 (27.96)

5. Other Pre Specified Outcome: Change in Clinician Administered PTSD Scale (CAPS) Score
Description: The CAPS is a 30-item structured interview that can be used to make current and lifetime diagnosis of post traumatic stress disorder (PTSD) as well as assess PTSD symptoms over the past week. Questions also examine the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS administration, overall response validity, overall PTSD severity, and specifications for the dissociative subtype (depersonalization and derealization). The identification of an index traumatic event to serves as the basis for symptom inquiry. The full interview takes approximately 45-60 minutes to administer. Items are scored from 0 to 4 where 0 = the symptom is absent and 4 = the symptom is incapacitating. A symptom severity score is obtained by summing items 1-20. Total scores range from 0 to 80 and a higher score indicates more severe PTSD symptoms.
Time Frame: Baseline
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Mini International Neuropsychiatric Interview (MINI) Score
Description: Mini International Neuropsychiatric Interview is a semistructured interview that will be used to assess for concurrent mood, substance, and psychotic disorders. The interview takes 30 minutes - 1 hour to administer. Participants answer "yes" or "no" to questions about symptoms they have been having; from these responses a clinician can diagnose lifetime and/or current presence of 22 psychiatric conditions. The number of instrument items used per interview depends on responses to previous questions and the interview is not designed to provide a numeric total score.
Time Frame: Baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Kreek-McHugh-Schluger-Kellogg (KMSK) Marijuana/Cannabis Scale Score
Description: This is a clinical measure designed to quickly assess the nature and extent of recreational use of cannabis during the last 24 hours. The instrument includes a 15-item scale where respondents indicate how much the agree with reasons for using marijuana, where 0 = strongly disagree and 5 = strongly agree. The full measure will be administered at the beginning of study participation, and one question about drug use in the past day (if applicable) will be administered on study intervention days.
Time Frame: Baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Affective Number Stroop (ANS) Task Score
Description: During the Affective Number Stroop (ANS) Task, participants are instructed to rapidly identify the number of numbers in a given display while ignoring evocative distractor images (trauma-relevant scenes) while in a MRI scanner. In these trials, the number of numbers presented is either consistent or inconsistent with the actual number displayed, such that there are both congruent and incongruent trials. The participants will be presented with positive and neutral pictures in addition to the negative trauma-relevant images. The task will be completed in the MRI scanner during both the pre- and post-treatment sessions.
Time Frame: Up to Week 4
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Penn Computerized Neuropsychological Battery Performance
Description: This is a computerized neuropsychological assessment that is designed to examine different domains of cognitive functioning. The executive functioning and memory components of this battery will be administered, which take approximately 30 minutes to complete.
Time Frame: Up to Week 4
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Posttraumatic Avoidance Behaviour Questionnaire (PABQ) Score
Description: The PABQ includes 25 items asking participants how often they engaged in certain behaviors in the past 3 weeks. Responses are given on a 4-point scale where 1 = almost never and 4 = almost always. Total scores range from 25 to 100 and higher scores indicate greater avoidance. This questionnaire will be given at post-treatment and follow-up time points to capture participants' avoidance behaviors during this time.
Time Frame: Week 4 (post-treatment), Week 8 (one month post-treatment)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Chesney's Coping Self-Efficacy Scale (CSES) Score
Description: The CSES is a 26-item scale that measures one's perceived ability to cope with life's difficulties. Responses are given on a scale from 0 to 10 where 0 = cannot do at all and 10 = certain can do. Total scores range from 0 to 260 where higher scores indicate greater self-efficacy with coping skills.
Time Frame: Baseline, Week 4 (post-treatment), Week 8 (one month post-treatment)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in State Self Efficacy Scale Score
Description: This is a 7 Item measure using a 7-point likert scale that will examine changes over time in self-efficacy on a state level. Responses to items range from 1 = strongly disagree to 7 = strongly agree. Total scores range from 1 to 49 where higher scores indicate greater self-efficacy.
Time Frame: Baseline, Week 4 (post-treatment), Week 8 (one month post-treatment)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Moral Injury Events Scale for Civilians (MIES-C) Score
Description: The Moral Injury Events Scale for Civilians (MIES-C) measurement is a 10-item scale assessing for the presence of potentially morally injurious events and feelings of distress that can emerge in the aftermath of these events. Responses are given on a 6-point scale where 1 = strongly agree and 6 = strongly disagree. Total scores range from 10 to 60 and lower scores indicate more exposure to events that conflict with the respondents sense of right and wrong.
Time Frame: Baseline
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Attentional Control Scale (ACS) Score
Description: This is a 20-item self-report measure that assesses attentional control a 4-point Likert scale, where 1 = almost never and 4 = always. Total scores range from 20 to 80 and higher scores indicate greater difficulty with attentional control.
Time Frame: Baseline, Week 4 (post-treatment), Week 8 (one month post-treatment)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in Difficulties in Emotion Regulation Scale (DERS)
Description: The DERS is a 36 item instrument that measures emotional dysregulation symptoms. Responses are given on a 5-point scale where 1 = almost never and 5 = almost always. The DERS scales include 1) nonacceptance of emotional responses, 2) difficulty engaging in goal-directed behavior, 3) difficulties with impulse control, 4) limited emotional awareness, 5) limited access to emotion regulation strategies, and 6) lack of emotional clarity. Total scores range from 36 to 180 and higher scores suggest greater problems with emotion regulation.
Time Frame: Baseline, Week 4 (post-treatment), Week 8 (one month post-treatment)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in State Trait Anxiety Inventory (STAI) Score
Description: The STAI is a 40-item self-report measure that uses a 4-point Likert scale to evaluate both state and trait anxiety. Total scores range from 40 to 160 and items are scored so that a higher total score indicates greater symptoms of anxiety. This is administered at the pre-MRI and post-MRI data collection points for every MRI visit.
Time Frame: Baseline up to Week 4 (post-treatment)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in Visual Analogue Scale (VAS) Score
Description: This is a 6-item self-report measure that indicates how intense one is feeling certain emotions using a 10-point Likert scale. Total scores range from 0 to 60 with higher scores indicating greater intensity of emotions.
Time Frame: Baseline, Week 4 (post-treatment)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change in Motivation and Pleasure -Self Report (MAP-SR) Score
Description: The MAP-SR is an 18-item self-report measure that assesses the motivation and pleasure domain of negative symptoms. Items are rated on a 5-point Likert scale and total scores range from 0 to 72. Certain items are reverse scored so that lower scores indicate greater pathology.
Time Frame: Baseline, Week 4 (post-treatment), Week 8 (one month post-treatment)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change in State Mindfulness Scale (SMS) Score
Description: This is a 21-item self-report measure that uses a 5-point Likert scale to assess one's perceived level of awareness and attention to the present moment and environment within a given frame of time (i.e. the last 10 minutes). This is administered before and after each intervention session. Responses are given on a scale from 1 (not at all) to 5 (very well). Total scores range from 21 to 105 and higher scores indicate greater mindfulness.
Time Frame: Pre-intervention and post-intervention of each session up to Week 4
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Client Satisfaction Questionnaire (CSQ)
Description: The CSQ is an 11-item self-report measure to assess how the intervention satisfied the participant's expectations and/or if it helped their daily lives in any way. The questionnaire contains a mix of scaled responses and open ended questions and there is not a summary score for this measurement.
Time Frame: Week 4 (post-treatment)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the One Month Post-treatment visit (up to 8 weeks).
Arm/Group | Breath-Focused Meditation | Breath-Focused Meditation Plus Physiological Feedback
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/38
Other Adverse Events (participants affected / at risk) | 0/27 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT02754557/Prot_SAP_000.pdf